CLINICAL TRIAL: NCT05517590
Title: Effect of Intravenous Tranexamic Acid Plus Intramyometrial Desmopressin on Blood Loss During Laparoscopic Myomectomy: Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Intravenous Tranexamic Acid and Intramyometrial Desmopressin Effect on Blood Loss During Laparoscopic Myomectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Esra Ozbasli, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ATADEK-2022/05-33
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Leiomyoma, Uterine; Intraoperative Blood Loss
Keywords: Leiomyoma; Laparoscopic myomectomy; Tranexamic acid; Blood loss; İntramyometrial desmopressin
MeSH Terms: conditions — Leiomyoma; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient, the surgeon and the assistant that will collect the data will be masked about the patient's study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid and group (Group I) (Active Comparator): In Group I, 1 gram of tranexamic acid will be diluted into 100 ml of saline solution and administered at a rate of 100 ml/hr 10 minutes before the skin incision time.
  Interventions: Drug: Tranexamic acid
- Saline group (Group II) (Placebo Comparator): Group II placebo will be administered to the control group, and 100 ml of saline solution will be administered at a rate of 100 ml/hr 10 minutes before the skin incision time.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tranexamic acid — 1 gram of tranexamic acid will be diluted into 100 ml of saline solution and administered at a rate of 100 ml/hr 10 minutes before the skin incision time.
  Other Names: Group I
  Arms: Tranexamic acid and group (Group I)
Drug: Saline — 100 ml of saline solution will be administered at a rate of 100 ml/hr 10 minutes before the skin incision time.
  Other Names: Group II
  Arms: Saline group (Group II)

SUMMARY:
To evaluate the effect of intravenous tranexamic acid plus intramyometrial desmopressin administration on perioperative blood loss and blood transfusion need in laparoscopic myomectomy operation.

DETAILED DESCRIPTION:
Although complication rates such as bleeding are observed to be low in surgeries performed by experienced surgeons, sometimes severe bleeding that may require emergency blood transfusion can be encountered during myomectomy operation. Therefore, various medical treatments such as vasopressin, misoprostol, ascorbic acid are still being sought to reduce the amount of intraoperative bleeding. Tranexamic acid is a lysine-derived drug with an antifibrinolytic effect, which has been used for a long time, especially in orthopedic and cardiovascular surgeries, to stop bleeding and reduce the need for blood transfusions, and is often well tolerated and has few side effects. It has a good safety profile with the Food and Drug Administration (FDA) Pregnancy Category B and is a drug frequently used in postpartum hemorrhage. It is also used to reduce bleeding in bleeding observed in many gynecological surgeries such as hypermenorrhea, bleeding in intrauterine device application and cervical conization. In the investigator's clinic, intramyometrial desmopressin administration is routinely used in most cases. Although the application of various intraoperative medical treatments in laparoscopic myomectomies has been examined in the literature, there are not enough prospective studies investigating the administration of desmopressin and intravenous tranexamic acid. In the investigator's study, investigators plan to evaluate the effect of the combined use of these two drugs on intraoperative bleeding and the need for blood transfusion compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer female patients over the age of 18 who will undergo laparoscopic myomectomy in our clinic will be included in our study.

Exclusion Criteria:

1. Patients who are planned to undergo different surgery along with myomectomy
2. Those with a diagnosis and suspicion of malignancy
3. Those with a history of thromboembolic disease
4. Those with cardiac, hepatic or renal disease
5. Those with a body mass index of 30 and above
6. Patients with abnormal coagulation test results
7. Patients using anticoagulants
8. Those who use drugs or diseases that may affect coagulation (serum creatinine > 1.5 mg/dL)
9. Those allergic to tranexamic acid

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss | At the end of the surgery.
  The amount of perioperative bleeding will be calculated by measuring the blood volume in the suction device and subtracting the irrigation fluid from the total amount.
Preoperative and postoperative hemoglobin change | On postoperative day 0 and day 2
  Preoperative and postoperative hemoglobin values will be recorded.

SECONDARY OUTCOMES:
Need for postoperative blood transfusion | Postoperative day 1
  Patients who received postoperative blood transfusions will be recorded.
Operation time | At the end of the operation.
  Operation time will be recorded.
Postoperative thrombosis symptoms | At postoperative first week and 3rd month.
  Postoperative thrombosis symptoms will be recorded at postoperative first week and 3rd month.

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, Study Director — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis might be shared when the study is completed upon request.

REFERENCES:
- [Background] Okolo S. Incidence, aetiology and epidemiology of uterine fibroids. Best Pract Res Clin Obstet Gynaecol. 2008 Aug;22(4):571-88. doi: 10.1016/j.bpobgyn.2008.04.002. Epub 2008 Jun 4. PMID 18534913
- [Background] Buckley VA, Nesbitt-Hawes EM, Atkinson P, Won HR, Deans R, Burton A, Lyons SD, Abbott JA. Laparoscopic myomectomy: clinical outcomes and comparative evidence. J Minim Invasive Gynecol. 2015 Jan;22(1):11-25. doi: 10.1016/j.jmig.2014.08.007. Epub 2014 Aug 10. PMID 25117840
- [Background] Jin C, Hu Y, Chen XC, Zheng FY, Lin F, Zhou K, Chen FD, Gu HZ. Laparoscopic versus open myomectomy--a meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2009 Jul;145(1):14-21. doi: 10.1016/j.ejogrb.2009.03.009. Epub 2009 Apr 23. PMID 19398260
- [Background] LaMorte AI, Lalwani S, Diamond MP. Morbidity associated with abdominal myomectomy. Obstet Gynecol. 1993 Dec;82(6):897-900. PMID 8233261
- [Background] Kongnyuy EJ, Wiysonge CS. Interventions to reduce haemorrhage during myomectomy for fibroids. Cochrane Database Syst Rev. 2014 Aug 15;2014(8):CD005355. doi: 10.1002/14651858.CD005355.pub5. PMID 25125317
- [Background] Opoku-Anane J, Vargas MV, Marfori CQ, Moawad G, Maasen MS, Robinson JK. Intraoperative tranexamic acid to decrease blood loss during myomectomy: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 2020 Sep;223(3):413.e1-413.e7. doi: 10.1016/j.ajog.2020.02.019. Epub 2020 Mar 28. PMID 32229194
- [Background] Srivastava S, Mahey R, Kachhawa G, Bhatla N, Upadhyay AD, Kriplani A. Comparison of intramyometrial vasopressin plus rectal misoprostol with intramyometrial vasopressin alone to decrease blood loss during laparoscopic myomectomy: Randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:279-283. doi: 10.1016/j.ejogrb.2018.07.006. Epub 2018 Jul 5. PMID 30056355
- [Background] Winkler UH. The effect of tranexamic acid on the quality of life of women with heavy menstrual bleeding. Eur J Obstet Gynecol Reprod Biol. 2001 Dec 1;99(2):238-43. doi: 10.1016/s0301-2115(01)00414-6. PMID 11788179